CLINICAL TRIAL: NCT07104344
Title: A Single-center, Open-label, Single-arm Clinical Study to Observe the Safety and Efficacy of CM355 in the Treatment of Refractory Systemic Lupus Erythematosus
Brief Title: Study of CM355 in Patients With Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM355_SLE_IIT
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CM355 (Experimental)
  Interventions: Biological: CM355

INTERVENTIONS:
Biological: CM355 — CM355 injection

SUMMARY:
This study was designed to investigate the safety and efficacy of CM355 in patients with refractory SLE.

DETAILED DESCRIPTION:
This study is designed to investigate the safety and efficacy of CM355 in patients with moderately to severely active SLE who are refractory to treatment, and to analyze its pharmacokinetic profile , pharmacodynamic effects, and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the nature of the study and voluntarily sign the informed consent form (ICF);
* Age ≥ 18 to ≤ 65 years old, male or female;
* At screening, patients must meet the 2019 European League Against Rheumatism (EULAR)/ American college of Rheumatology (ACR)classification criteria for systemic lupus erythematosus (SLE) as assessed by a qualified doctor, and have a disease course of ≥ 12 months；
* systemic lupus erythematosus disease activity index2000 (SLEDAI-2K)≥8 points at screening. If there is a low complement and/or anti-ds-DNA antibody score, the SLEDAI-2K) clinical symptoms (excluding low complement and/or anti-ds-DNA antibody) score ≥ 6 points or ≥ 1 organ system in BILAG score should be Class A at screening；
* Definition of refractory SLE;
* The treatment regimen for SLE was stable for more than 4 weeks before the first dose.

Exclusion Criteria:

* Renal disease: patients with severe lupus nephritis;
* Patients with central nervous system diseases;
* Patients who have received monoclonal antibodies targeting Cluster of Differentiation 19(CD19) or Cluster of Differentiation 20(CD20) or other B-cell depleting agents within 6months prior to the first dose ;
* Any other condition assessed by investigator as unsuitable for participation in the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
adverse events (AE) | Throughout the study，an average of about 1 year
  Incidence and severity of adverse events (AE)

CONTACTS AND LOCATIONS:
Overall Officials: Hai Long, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No